CLINICAL TRIAL: NCT05525962
Title: Facteurs de vulnérabilité/résilience influençant Les Trajectoires développementales et Les modalités Adaptatives d'Enfants et d'Adolescents confiés à l'Aide Sociale à l'Enfance. Cohorte Primo-arrivants.
Brief Title: Vulnerability/Resilience Factors Influencing the Developmental Trajectories and Adaptive Methods of Children and Adolescents in Child Welfare System.
Acronym: EvolASE-PEA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0219/HP
Record Dates: First submitted 2022-06-23; First posted 2022-09-02 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Behavior, Child; Child Development; Child Development Disorder; Adolescent Development; Adolescent Behavior; Child Mental Disorder; Child Behavior Disorders; Adolescent - Emotional Problem
Keywords: child; preschool; adolescent; psychiatry; psychology; Child Protective Services; social sciences; child protection; social services; psychiatric disorders; attachement; developmental trajectories
MeSH Terms: conditions — Child Behavior; Developmental Disabilities; Adolescent Behavior; Neurodevelopmental Disorders; Child Behavior Disorders; Mental Disorders | interventions — Weights and Measures; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: questionnaries, scales, cognitive tests — A first interview is planned with a psycholgist in the weeks following the minor arrival in the structure (M0)
  * M0: cognitive test, psychiatric classification and psychologic assessments
  * M12 and M24: psychiatric classification and psychologic assessments

SUMMARY:
Assess the prevalence of medico-psychological characteristics at the time of placement (M0), their appearance / disappearance and during the two years following placement (M12 and M24) by age group in children / adolescents in Child Protective Services and placed full-time in the structures of Seine-Maritime and Eure as well as in nursery in Le Havre or Rouen

ELIGIBILITY:
Inclusion Criteria:

* Minor adressed to child protective services
* Minor placed full time

Exclusion Criteria:

* Non affiliation to social security system
* Non accompanied minor
* Minor and/or parfents not understanding french
* Minor informed and refused participation
* Parents or tutor having refused participation of their child

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Minor (0 to 16 years old) arriving for the first time in child protective system and present full time
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Presence and nature of psychiatric disorders according to DSM 5 | At inclusion
  assessed by MINI S-KID (International Neuropsychiatric Interview for Children and Adolescents) for 6-18 year olds and DC 0-5 (Diagnostic Classification from 0 to 5 ) for 0 to 5 year olds.
Presence and nature of psychiatric disorders according to DSM 5 | 1 year after inclusion
  assessed by MINI S-KID (International Neuropsychiatric Interview for Children and Adolescents) for 6-18 year olds and DC 0-5 (Diagnostic Classification from 0 to 5 ) for 0 to 5 year olds.
Presence and nature of psychiatric disorders according to DSM 5 | After 2 years
  assessed by MINI S-KID (International Neuropsychiatric Interview for Children and Adolescents) for 6-18 year olds and DC 0-5 (Diagnostic Classification from 0 to 5 ) for 0 to 5 year olds.

SECONDARY OUTCOMES:
Description of cognitive abilities | At inclusion
  0 to 2 years old : BAYLEY V3 or Brunet Lezine (revised) 3 to 6 years old : WPPSI-IV 7 to 16 years old : WISC-V 16 to 18 years old : WAIS-V
Presence of an attachement psychopathological disorder | At inclusion
  Assessed by the strange situation procedure for participants aged from 9 months old to 3 years old Assessed by Attachment story completion test from 4 to 9 years old Assessed by the Inventory of Parents and Peer Attachement from 10 to 18 years old
Presence of a Borderline-Personality-Disorder | At inclusion
  Using AbDIB questionnaire from 12 to 18 years old
Presence of an emotional and behavioral; self-regulation Disorder | At inclusion
  - 1.5 -18 ans : Child Behavior Checklist (CBCL)
Presence of an emotional and behavioral; self-regulation Disorder | At inclusion
  - 6-18 ans : Affective Reactivity Index Child Report and Parent Report (ARI)
Presence of an emotional and behavioral; self-regulation Disorder | At inclusion
  - 9-18 ans: Toronto Alexithymia Scale (TAS-20)
Presence of an emotional and behavioral; self-regulation Disorder | At inclusion
  - 6-18 ans : Rosenberg self-assessment scale - (RSE)
Presence of one or multisensory hallucinations | At inclusion
  6 -18 ans: Multisensory Hallucinations Scale for Children (MHASC)
Mentalization capacities | At inclusion
  12 to 18 using the Reflective Functioning Questionnaire (RFQ 20)
Presence of eating disorder | At inclusion
  2 -18 : SCOFF questionnaire
Substance use disorders | At inclusion
  11 to 18 years old using the Detection of alcohol and drugs problems in adolescent (DepAdo)
Analyses of adverse life events | At inclusion
  - UCLA Child/Adolescent PTSD Reaction Index (PTSD-UCLA)
Analyses of adverse life events | At inclusion
  - 11 - 18 years old: Childhood Trauma Questionnaire (CTQ)
Description of care pathway | At inclusion
  using a socio-demographic report (scolarship, medical care and environnement)
Coping strategies | At inclusion
  - 12 to 18 years old using the Adolescent Coping Scale (ACS)
Coping strategies | At inclusion
  - 7 to 13 years old : Self-Report Coping Scale (SRCS)
Coping strategies | After 1 year
  - 12 to 18 years old using the Adolescent Coping Scale (ACS)
Coping strategies | After 1 year
  - 7 to 13 years old : Self-Report Coping Scale (SRCS)
Coping strategies | After 2 years
  - 12 to 18 years old using the Adolescent Coping Scale (ACS)
Coping strategies | After 2 years
  - 7 to 13 years old : Self-Report Coping Scale (SRCS)
Presence of depressive symptoms | At inclusion
  12-18 years old: Columbia-Suicide Severity Rating Scale (C-SSRS)
Analyses of global functionning | At inclusion
  Using the global assessment functionning
Analyses of global functionning | At inclusion
  Using Ages & Stages Questionnaires Version 3 (ASQ3)
Presence of attachement psychopathological disorder | 1 year after inclusion
  Assessed by the strange situation procedure for participants aged from 9 months old to 3 years old Assessed by Attachment story completion test from 4 to 9 years old Assessed by the Inventory of Parents and Peer Attachement from 10 to 18 years old
Presence of a Borderline-Personality-Disorder | After 1 year
  Using AbDIB questionnaire from 12 to 18 years old
Presence of Emotional and behavioral, self-regulation Disorder | 1 year after inclusion
  - 1.5 -18 ans : Child Behavior Checklist (CBCL)
Presence of Emotional and behavioral, self-regulation Disorder | 1 year after inclusion
  - 6-18 ans : Affective Reactivity Index Child Report and Parent Report (ARI)
Presence of Emotional and behavioral, self-regulation Disorder | 1 year after inclusion
  - 9-18 ans: Toronto Alexithymia Scale (TAS-20)
Presence of Emotional and behavioral, self-regulation Disorder | 1 year after inclusion
  - 6-18 ans : Rosenberg self-assessment scale - (RSE)
Presence of one or multisensory hallucinations | 1 year after inclusion
  6 -18 ans: Multisensory Hallucinations Scale for Children (MHASC)
Mentalization capacities | 1 year after inclusion
  12 to 18 years old using the Reflective Functioning Questionnaire (RFQ 20)
Presence of eating disorder | 1 year after inclusion
  2 -18 : SCOFF questionnaire
Substance use disorders | 1 year after inclusion
  11 to 18 years old using the Detection of alcohol and drugs problems in adolescent (DepAdo)
Analyses of adverse life events | 1 year after inclusion
  - UCLA Child/Adolescent PTSD Reaction Index (PTSD-UCLA)
Analyses of adverse life events | 1 year after inclusion
  - 11 - 18 years old: Childhood Trauma Questionnaire (CTQ)
Description of care pathway | 1 year after inclusion
  using a socio-demographic report (scolarship, medical care and environnement)
Presence of depressive symptoms | 1 year after inclusion
  12-18 years old: Columbia-Suicide Severity Rating Scale (C-SSRS)
Analyses of global functionning | 1 year after inclusion
  Using the global assessment functionning and the Ages & Stages Questionnaires Version 3 (ASQ3)
Presence of a attachement psychopathological disorder | 2 years after inclusion
  Assessed by the strange situation procedure for participants aged from 9 months old to 3 years old Assessed by Attachment story completion test from 4 to 9 years old Assessed by the Inventory of Parents and Peer Attachement from 10 to 18 years old
Presence of a Borderline-Personality-Disorder | 2 years after inclusion
  Using AbDIB questionnaire from 12 to 18 years old
Presence of a Emotional and behavioral self-regulation Disorder | 2 years after inclusion
  - 1.5 -18 ans : Child Behavior Checklist (CBCL)
Presence of a Emotional and behavioral self-regulation Disorder | 2 years after inclusion
  - 6-18 ans : Affective Reactivity Index Child Report and Parent Report (ARI)
Presence of a Emotional and behavioral self-regulation Disorder | 2 years after inclusion
  - 9-18 ans: Toronto Alexithymia Scale (TAS-20)
Presence of a Emotional and behavioral self-regulation Disorder | 2 years after inclusion
  - 6-18 ans : Rosenberg self-assessment scale - (RSE)
Presence of one or multisensory hallucinations | 2 years after inclusion
  - 6 -18 ans: Multisensory Hallucinations Scale for Children (MHASC)
Mentalization capacities | 2 years after inclusion
  12 to 18 years old using the Reflective Functioning Questionnaire (RFQ 20)
Presence of eating disorder | 2 years after inclusion
  2 -18 : SCOFF questionnaire
Substance use disorders | 2 years after inclusion
  11 to 18 years old using the Detection of alcohol and drugs problems in adolescent (DepAdo)
Analyses of adverse life events | 2 years after inclusion
  - UCLA Child/Adolescent PTSD Reaction Index (PTSD-UCLA)
Analyses of adverse life events | 2 years after inclusion
  - 11 - 18 years old: Childhood Trauma Questionnaire (CTQ)
Analyses of global functionning | 2 years after inclusion
  Using the global assessment functionning
Analyses of global functionning | 2 years after inclusion
  Using the Ages & Stages Questionnaires Version 3 (ASQ3)
Description of care pathway | 2 years after inclusion
  using a socio-demographic report (scolarship, medical care and environnement)
Presence of depressive symptoms | 2 years after inclusion
  12-18 years old: Columbia-Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - IDEFHI, Canteleu
  - Foyer Départementale de l'Enfance, Évreux
  - Centre infantile Raymond Lerch, Le Havre
  - Centre hospitalier du Belvédère, Mont-Saint-Aignan
  - Fondation les Nids, Mont-Saint-Aignan